CLINICAL TRIAL: NCT04371302
Title: Nursing Perspective on Burnout and Medical Errors in the Intensive Care Unit of an Exclusively Covid-19 Hospital: the Malaysian Experience
Brief Title: Nursing Perspective on Burnout and Medical Errors in the Intensive Care Unit During Covid-19 Pandemic
Status: Terminated | Type: Observational
Why Stopped: Logistical problems, administrative issues
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Samuel E H Tsan, MD, BMedSc, Doctor, University of Malaya
Other Study IDs: 54843
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Burnout, Professional; Medical Errors; Depression
Keywords: Burnout; Depression; Medical errors; Intensive Care Unit nurses; Covid-19
MeSH Terms: conditions — Burnout, Professional; Depression; Burnout, Psychological; COVID-19 | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive Care Unit nurses: Nurses working in the Intensive care Unit of an exclusive Covid-19 hospital in Malaysia, during the Covid-19 pandemic
  Interventions: Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Questionnaire — Assessment of demographics, burnout, depression and self-perceived medical errors

SUMMARY:
The investigators plan to perform an observational study to evaluate the prevalence of burnout, depression and medical errors in a designated exclusive Covid-19 patients hospital in Malaysia, during the Covid-19 pandemic. In addition, the relationship between burnout and depression with medical errors will be assessed. The population studied will be the nurses working in the Intensive Care Unit, who are at higher risk due to the nature of their work at the frontlines of the pandemic.

DETAILED DESCRIPTION:
During this unprecedented Covid-19 pandemic crisis in the whole world, Malaysia is also affected, with more than 5000 patients infected in the whole country as of 20th April, 2020. Many Intensive Care Unit nurses, who are at the frontlines of managing Covid-19 patients, face increased workload, in addition to psychological stress from managing these patients, with stress also coming from being exposed to the risk of cross infection. Hence, they are possibly at high risk of burnout and depression. In such a time of increased stress, the investigators also seek to find out the prevalence of medical errors made by Intensive Care Unit nurses during this pandemic, and whether the medical errors are associated with burnout. Factors associated with burnout, depression and medical errors will also be evaluated.

ELIGIBILITY:
Inclusion criteria

1. All nurses currently serving in the ICU, Sungai Buloh Hospital

Exclusion criteria

1. Subjects who refuse to participate
2. Subjects working in ICU, Sungai Buloh Hospital, for less than 1 month

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All ICU nurses serving in Sungai Buloh Hospital, a nationally designated exclusive Covid-19 hospital in Malaysia during the Covid-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of burnout among ICU nurses during Covid-19 | 2 months
  Prevalence of burnout risk
Prevalence of depression among ICU nurses during Covid-19 | 2 months
  Prevalence of depression risk
Prevalence of self-perceived medical errors among ICU nurses during Covid-19 | 2 months
  Prevalence of self perceived medical errors
Association of burnout, depression and medical errors among anaesthesiology clinicians during Covid-19 | 2 months
  To find out if there exists a relationship between burnout, depression and medical errors

CONTACTS AND LOCATIONS:
Locations (1):
- Sungai Buloh Hospital, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No